CLINICAL TRIAL: NCT00717067
Title: An Open-Label, Parallel Group, Single And Multiple Dose Study To Evaluate The Pharmacokinetics, Safety And Toleration Of Maraviroc Administered To Subjects With Various Degrees Of Renal Impaired And Normal Renal Function
Brief Title: Pharmacokinetics, Safety And Toleration Of Maraviroc Administered To Subjects With Various Degrees Of Renal Impaired And Normal Renal Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4001075
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Results first posted 2009-12-21 (Estimated); Last update posted 2010-11-19 (Estimated); Status verified 2010-11

CONDITIONS: Human Immunodeficiency Virus (HIV) Infection
Keywords: maraviroc, pharmacokinetics, renal impairment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Renal Insufficiency | interventions — Maraviroc; Ritonavir; Saquinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Healthy Subjects (Experimental): Subjects with Normal Renal Function (Creatinine Clearance > 80mL/min) (I) Maraviroc single dose, followed by (II) Maraviroc + Saquinavir/Ritonavir
  Interventions: Drug: Maraviroc; Drug: Ritonavir; Drug: Saquinavir
- Mild Renal Impairment (Experimental): Subjects with Mild Renal Impairment (Creatinine Clearance >50 and ≤80 mL/min)
  Interventions: Drug: Maraviroc; Drug: Ritonavir; Drug: Saquinavir
- Moderate Renal Impairment (Experimental): Subjects with Moderate Renal Impairment (Creatinine Clearance ≥30 and ≤50 mL/min)
  Interventions: Drug: Maraviroc; Drug: Ritonavir; Drug: Saquinavir
- Severe Renal Impairment (Experimental): Subjects with Severe Renal Impairment (Creatinine Clearance <30 mL/min)
  Interventions: Drug: Maraviroc
- ESRD on Hemodialysis (Experimental): Subjects with End Stage Renal Impairment receiving Hemodialysis(Creatinine Clearance <30 mL/min) (I) Maraviroc single dose one hour following completion of hemodialysis, followed by (II) Maraviroc single dose three hours prior to start of hemodialysis
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc 300 mg (150 mg x 2 tablets) x single dose
  Arms: Healthy Subjects
Drug: Maraviroc — Maraviroc 150 mg tablet twice daily x 7 days
  Arms: Healthy Subjects
Drug: Ritonavir — Ritonavir 100 mg capsule twice daily x 7 days
  Arms: Healthy Subjects
Drug: Saquinavir — Saquinavir 1000 mg (500 mg x 2 tablets) twice daily x 7 days
  Arms: Healthy Subjects
Drug: Maraviroc — Maraviroc 150 mg tablet once daily x 7 days
  Arms: Mild Renal Impairment
Drug: Ritonavir — Ritonavir 100 mg capsule twice daily x 7 days
  Arms: Mild Renal Impairment
Drug: Saquinavir — Saquinavir 1000 mg (500 mg x 2 tablets) twice daily x 7 days
  Arms: Mild Renal Impairment
Drug: Maraviroc — Maraviroc 150 mg tablet once every 48 hours x 7 days
  Arms: Moderate Renal Impairment
Drug: Ritonavir — Ritonavir 100 mg capsule twice daily x 7 days
  Arms: Moderate Renal Impairment
Drug: Saquinavir — Saquinavir 1000 mg (500 mg x 2 tablets) twice daily x 7 days
  Arms: Moderate Renal Impairment
Drug: Maraviroc — Maraviroc 300 mg (150 mg x 2 tablets) x single dose
  Arms: Severe Renal Impairment
Drug: Maraviroc — Maraviroc 300 mg (150 mg x 2 tablets) x single dose one hour following completion of hemodialysis
  Arms: ESRD on Hemodialysis
Drug: Maraviroc — Maraviroc 300 mg (150 mg x 2 tablets) x single dose three hours prior to start of hemodialysis
  Arms: ESRD on Hemodialysis

SUMMARY:
The purpose of this study is to assess whether a dosing adjustment is needed in patients with renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Stable Renal Function defined as ≤20% (25% for normal renal function) difference between 2 measurements of serum creatinine obtained on 2 occasions separated by at least 2 weeks.
* Body Mass Index (BMI) of approximately 18 to 40 kg/m2 inclusive.
* Total body weight >50 kg (110 lbs).
* Male or female subjects between the ages of 18 and 85 years.

Exclusion Criteria:

* Subjects with acute renal disease and/or history of renal transplant.
* Supine BP at Screening ≥160 mm Hg systolic or ≥95 mm Hg diastolic.
* Supine BP at Screening ≤80 mm Hg systolic or ≤40 mm Hg diastolic.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Germany (2):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, München

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001075&StudyName=Pharmacokinetics%2C%20Safety%20And%20Toleration%20Of%0AMaraviroc%20Administered%20To%20Subjects%20With%20Various%20Degrees%20Of%20Renal%20Impaired%20And%20Normal%20Renal%20Fu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two centers took part in this study between 15 July 2008 and 21 November 2008.
Pre-assignment Details: Subjects were enrolled into treatment groups (healthy subjects, mild, moderate, severe renal impairment, or end stage renal impairment on hemodialysis) based on creatinine clearance results obtained closest to the dosing date at screening as determined by the Cockcroft-Gault equation (with the exception of subjects undergoing hemodialysis).
Groups:
- Healthy Subjects: (I) Maraviroc single 300 mg dose, followed 4 days later by (II) Maraviroc 150 mg twice a day (BID) co-administered with saquinavir 1,000 mg/ritonavir 100 mg twice a day (BID) for 6 days, and a single dose of both agents on Day 7.
- Mild Renal Impairment: Maraviroc 150 mg once a day (QD) co-administered with saquinavir 1,000 mg/ritonavir 100 mg twice a day (BID) for 7 days.
- Moderate Renal Impairment: Maraviroc 150 mg every 48 hours co-administered with saquinavir 1,000 mg/ritonavir 100 mg twice a day (BID) for 7 days.
- Severe Renal Impairment: Maraviroc 300 mg single dose.
- ESRD: Single Dose: (I) Maraviroc single dose one hour following completion of morning hemodialysis, followed at least 1 week later by (II) Maraviroc single dose three hours prior to start of hemodialysis.
Period: Part 1a: Normal/Mild/Moderate Group
Arm/Group | Healthy Subjects | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | ESRD: Single Dose
Started | 6 | 6 | 6 | 0 | 0
Completed | 6 | 6 | 5 | 0 | 0
Not Completed | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Period: Part 1b: Severe Renal Impairment
Arm/Group | Healthy Subjects | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | ESRD: Single Dose
Started | 0 | 0 | 0 | 6 | 0
Completed | 0 | 0 | 0 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Part 2: End Stage Renal Disease
Arm/Group | Healthy Subjects | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | ESRD: Single Dose
Started | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Subjects: Subjects with Normal Renal Function (Creatinine Clearance > 80mL/min)
- ESRD on Hemodialysis: Subjects with End Stage Renal Disease Requiring Regular Hemodialysis 3 Times a Week for at Least 6 Weeks Prior to Screening (Creatinine Clearance <30 mL/min)
- Total: Total of all reporting groups
Arm/Group | Healthy Subjects | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | ESRD on Hemodialysis | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 30
Age, Customized [Number; unit: years]
  18 - 44 years | 0 | 0 | 1 | 1 | 1 | 3
  45 - 64 years | 5 | 4 | 0 | 2 | 4 | 15
  >= 65 years | 1 | 2 | 5 | 3 | 1 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 0 | 8
  Male | 4 | 4 | 4 | 4 | 6 | 22

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time-curve From Zero to the Last Measured Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast) measured in nanograms * hour divided by milliliters (ng*hr/mL).
Time Frame: Pre-dose, post-dose hours 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72.
Population: Pharmacokinetic (PK) parameter analysis population: all subjects treated who have at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Healthy Subjects: Multiple Dose: Maraviroc 150 mg twice a day (BID) co-administered with saquinavir 1,000 mg/ritonavir 100 mg twice a day (BID) for 6 days, and a single dose of both agents on Day 7.
- Mild Renal Impairment: Multiple Dose: Maraviroc 150 mg once a day (QD) co-administered with saquinavir 1,000 mg/ritonavir 100 mg twice a day (BID) for 7 days.
- Moderate Renal Impairment: Multiple Dose: Maraviroc 150 mg every 48 hours co-administered with saquinavir 1,000 mg/ritonavir 100 mg twice a day (BID) for 7 days.
- Healthy Subjects: Single Dose; Severe Renal Impairment: Single Dose: Maraviroc 300 mg single dose.
- ESRD: Single Dose; After Dialysis: Maraviroc 300 mg single dose one hour following completion of morning hemodialysis.
- ESRD: Single Dose; Before Dialysis: Maraviroc 300 mg single dose three hours prior to start of hemodialysis.
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose | ESRD: Single Dose; After Dialysis | ESRD: Single Dose; Before Dialysis
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6
ng*hr/mL | 7356.3 (2313.45) | 9502.1 (3599.32) | 6496.0 (1795.89) | 1320.7 (988.66) | 4255.5 (2424.19) | 2636.5 (1123.34) | 2770.1 (1356.56)
Statistical Analysis 1: Comparison: Healthy Subjects: Multiple Dose vs Mild Renal Impairment: Multiple Dose; Ratio (%) test (mild) / reference (normal). AUClast was calculated using the log-linear trapezoidal method; Test type: Superiority or Other; ANOVA; ratio of adjusted geometric means = 129.17, 90% CI [92.16 to 181.04]
Statistical Analysis 2: Comparison: Healthy Subjects: Multiple Dose vs Moderate Renal Impairment: Multiple Dose; Ratio (%) test (moderate) / reference (normal). AUClast was calculated using the log-linear trapezoidal method; Test type: Superiority or Other; ANOVA; ratio of adjusted geometric means = 88.31, 90% CI [61.97 to 125.83]
Statistical Analysis 3: Comparison: Healthy Subjects: Single Dose vs Severe Renal Impairment: Single Dose; Ratio (%) test (severe) / reference (normal). AUClast was calculated using the log-linear trapezoidal method; Test type: Superiority or Other; ANOVA; ratio of adjusted geometric means = 322.23, 90% CI [171.97 to 603.78]

2. Primary Outcome: AUCtau
Description: AUCtau: area under the plasma concentration-time profile from time zero to the end of the dosing interval (tau); measured in nanograms * hours divided by milliliters (ng.hr/mL).
Time Frame: Pre-dose, post-dose hours 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72.
Population: Pharmacokinetic (PK) parameter analysis population: all subjects treated who have at least 1 of the PK parameters of interest. AUCtau for end stage renal disease subjects was not determined.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose
Number analyzed (Participants) | 6 | 6 | 5
ng*hr/mL | 5341.4 (1498.27) | 8118.7 (2995.27) | 6193.3 (1762.41)
Statistical Analysis 1: Comparison: Healthy Subjects: Multiple Dose vs Mild Renal Impairment: Multiple Dose; Ratio (%) test (mild) / reference (normal); Test type: Superiority or Other; ANOVA; ratio of adjusted geometric means = 151.99, 90% CI [109.53 to 210.92]
Statistical Analysis 2: Comparison: Healthy Subjects: Multiple Dose vs Moderate Renal Impairment: Multiple Dose; Ratio (%) test (moderate) / reference (normal); Test type: Superiority or Other; ANOVA; ratio of adjusted geometric means = 115.95, 90% CI [82.23 to 163.50]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax) within the dosing interval; measured in nanograms per milliliter (ng/mL).
Time Frame: Pre-dose, post-dose hours 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72.
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose | ESRD: Single Dose; After Dialysis | ESRD: Single Dose; Before Dialysis
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6
ng/mL | 950.91 (220.368) | 1150.74 (392.167) | 674.20 (275.722) | 335.60 (393.024) | 801.16 (525.656) | 576.7 (339.27) | 478.5 (198.81)
Statistical Analysis 1: Comparison: Healthy Subjects: Multiple Dose vs Mild Renal Impairment: Multiple Dose; Ratio (%) test (mild) / reference (normal); Test type: Superiority or Other; ANOVA; ratio of adjusted geometric means = 121.01, 90% CI [83.15 to 176.13]
Statistical Analysis 2: Comparison: Healthy Subjects: Multiple Dose vs Moderate Renal Impairment: Multiple Dose; Ratio (%) test (moderate) / reference (normal); Test type: Superiority or Other; ANOVA; ratio of adjusted geometric means = 70.90, 90% CI [47.83 to 105.10]
Statistical Analysis 3: Comparison: Healthy Subjects: Single Dose vs Severe Renal Impairment: Single Dose; Ratio (%) test (severe) / reference (normal); Test type: Superiority or Other; ANOVA; ratio of adjusted geometric means = 238.73, 90% CI [106.83 to 533.48]

4. Secondary Outcome: Plasma Protein Binding
Description: Percent protein binding (protein unbound maraviroc (MVC) fraction [percent free]) was determined by rapid equilibrium dialysis. Percent free = 100 - percent bound.
Time Frame: 2 hours post-dose; normal Day -3 and Day 7; mild moderate: Day 7; severe and ESRD: Day 1
Population: as for outcome 1
Measure: Number; unit: percent free
Groups:
- ESRD: (I) Maraviroc 300 mg single dose one hour following completion of morning hemodialysis, followed at least 1 week later by (II) Maraviroc 300 mg single dose three hours prior to start of hemodialysis.
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose | ESRD
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6
percent free
  minimum protein unbound MVC fraction | 19.7 [14.6 to 28.2] | 15.3 [15.3 to 29.1] | 18.1 [18.1 to 31.6] | 14.6 [19.2 to 28.1] | 19.2 [18.2 to 27.8] | 18.2 [18.2 to 27.8]
  maximum protein unbound MVC fraction | 26.6 | 29.1 | 31.6 | 28.2 | 28.1 | 27.8

5. Secondary Outcome: Area Under the Time Curve From 0 to Infinity (AUCinf)
Description: Area under the plasma concentration-time profile from time zero to the time infinate in subjects who received single dose treatment; measured in nanograms * hour divided by millilters (ng*hr/mL).
Time Frame: Pre-dose, post-dose hours 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72
Population: Pharmacokinetic (PK) parameter analysis population: all subjects treated who have at least 1 of the PK parameters of interest. AUC infinity was not determined for subjects in the multiple dose treatment groups.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose | ESRD: Single Dose; After Dialysis | ESRD: Single Dose; Before Dialysis
Number analyzed (Participants) | 6 | 6 | 6 | 6
ng*hr/mL | 1348.4 (986.65) | 4367.7 (2518.78) | 2677.4 (1149.85) | 2805.5 (1374.71)
Statistical Analysis 1: Comparison: Healthy Subjects: Single Dose vs Severe Renal Impairment: Single Dose; Ratio (%) test (severe) / reference (normal); Test type: Superiority or Other; ANOVA; ratio of adjusted geometric means = 323.91, 90% CI [174.32 to 601.88]

6. Secondary Outcome: Time of First Occurrence (Tmax)
Description: Time (hours) of first occurrence (Tmax); time after dosing when Cmax (maximum plasma concentration) occured.
Time Frame: Pre-dose, post-dose hours 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72.
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose | ESRD: Single Dose; After Dialysis | ESRD: Single Dose; Before Dialysis
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6
hours | 1.000 [0.50 to 2.00] | 1.500 [0.50 to 4.00] | 2.000 [0.50 to 4.02] | 2.500 [0.50 to 4.02] | 2.500 [0.50 to 4.00] | 3.000 [1.00 to 4.00] | 2.000 [0.50 to 4.17]

7. Secondary Outcome: Half-life (t1/2)
Description: Elimination half-life (t1/2) measured in hours: time required for half the quantity of maraviroc to be metabolized or eliminated by normal biological processes.
Time Frame: Pre-dose, post-dose hours 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose | ESRD: Single Dose; After Dialysis | ESRD: Single Dose; Before Dialysis
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6
hour | 14.22 (1.166) | 16.84 (5.568) | 16.99 (3.141) | 14.36 (4.030) | 17.29 (4.171) | 15.03 (3.329) | 13.86 (1.051)

8. Secondary Outcome: Renal Clearance (CLR) in Subjects With Normal, Mild, Moderate and Severe Renal Function
Description: Renal clearance (CLR) measured in milliliters per minute (mL/min).
Time Frame: Hour 0 (prior to MVC dosing [single dose] or prior to last MVC dose [multiple dose]) to 72 hours post-dose ; hours 0, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72.
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: mL/min
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
mL/min | 105.7 (56.00) | 77.2 (36.71) | 62.5 (12.57) | 110.0 (38.67) | 26.6 (18.84)

9. Secondary Outcome: Derivation of Renal Clearance in Subjects With Normal, Mild, Moderate and Severe Renal Function: Ae
Description: Ae: amount of drug excreted unchanged in the urine; measured in milligrams (mg).
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6
mg | 41.6 (22.45) | 39.1 (11.23) | 24.9 (8.88) | 10.8 (7.41) | 8.4 (6.35)

10. Secondary Outcome: Hemodialysis Clearance of Maraviroc (MVC) in Subjects With End Stage Renal Disease (ESRD) Undergoing Hemodialysis: CLdD
Description: CLdD: dialysate clearance before dialysis; measured in milliliters per minute.
Time Frame: Before dialysis
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: mL/min
Arm/Group | ESRD: Single Dose; Before Dialysis
Number analyzed (Participants) | 6
mL/min | 36.42 (12.710)

11. Secondary Outcome: Safety and Tolerability of Maraviroc in the Absence and Presence of a Potent CYP3A4 Inhibitor in Subjects With Various Degrees of Renal Impairment or Undergoing Hemodialysis: Number of Subjects With Maximum Increase and Decrease in Supine Blood Pressure
Description: Number of subjects with absolute values of supine systolic blood pressure (BP) measured in millimeters of mercury (mm/Hg), range: <90 mmHg; and supine diastolic blood pressure, range: <50 mmHg. Number of subjects with a maximum increase and decrease from Baseline in supine systolic BP ≥ 30 mmHg. Number of subjects with a maximum increase and decrease from Baseline in supine diastolic BP ≥ 20 mmHg.
Time Frame: Normal renal function: screening, Day -3 to Day -1; normal, mild and moderate RI: Day 7 to Day 10 and follow-up; severe RI: Day 1 to Day 4 and follow-up; ESRD: Day 1, Day 4, and follow-up
Population: Safety analysis set: all subjects who received study medication. BL: Baseline.
Measure: Number; unit: subjects
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose | ESRD: Single Dose; After Dialysis | ESRD: Single Dose; Before Dialysis
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6
subjects
  BL Supine Systolic Blood Pressure (BP) <90 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum Increase from BL: Supine Systolic BP≥ 30 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum Decrease from BL: Supine Systolic BP ≥ 30 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  BL Supine Diastolic Blood Pressure (BP) <50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum Increase from BL: Supine Diastolic BP≥ 20 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Maximun Decrease from BL: Supine Diastolic BP ≥20 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Safety and Tolerability of Maraviroc in the Absence and Presence of a Potent CYP3A4 Inhibitor in Subjects With Various Degrees of Renal Impairment or Undergoing Hemodialysis: Number of Subjects With Pulse Rate < 40 and > 120 Beats Per Minute
Description: Number of subjects with pulse rate < 40 beats per minute (BPM), number of subjects with pulse rate > 120 BPM.
Time Frame: as for outcome 11
Population: Safety analysis set: all subjects who received study medication.
Measure: Number; unit: bpm
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose | ESRD: Single Dose; After Dialysis | ESRD: Single Dose; Before Dialysis
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6
bpm
  Supine Pulse Rate <40 BPM | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine Pulse Rate >120 BPM | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Safety and Tolerability of Maraviroc in the Absence and Presence of a Potent CYP3A4 Inhibitor in Subjects With Various Degrees of Renal Impairment or Undergoing Hemodialysis: Number of Subjects With Maximum EGC QTC, QTCB and QTCF Intervals
Description: Single 12-lead ECG: number of subjects with maximum QTC interval, maximum QTCB interval (Bazett's correction), and maximum QTCF interval (Friderica's correction) measured in milliseconds (msec); range: 450 to <480 msec, 480 to <500 msec, and >500 msec. Maximum QTC interval increase from Baseline; citeria: change = ≥ 30 msec to < 60 msec, and change = ≥ 60 msec.
Time Frame: Normal renal function: screening, Day -3 and Day -1; normal renal function, mild and moderate RI: Day 7 to Day 9 and follow-up; severe RI: screening, Day 1, Day 3, Day 4, and follow-up; ESRD: screening, Day 1, Day 3, Day 4, and follow-up
Population: Safety analysis set: all subjects who received study medication.
Measure: Number; unit: subjects
Arm/Group | Healthy Subjects: Multiple Dose | Mild Renal Impairment: Multiple Dose | Moderate Renal Impairment: Multiple Dose | Healthy Subjects: Single Dose | Severe Renal Impairment: Single Dose | ESRD: Single Dose; After Dialysis | ESRD: Single Dose; Before Dialysis
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 6 | 6 | 6
subjects
  Maximum QTC Interval: 450 to < 480 msec | 1 | 0 | 0 | 1 | 2 | 1 | 0
  Maximum QTC Interval: 480 to < 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QTC Interval: > 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QTCB Interval: 450 to < 480 msec | 1 | 0 | 0 | 1 | 1 | 0 | 0
  Maximum QTCB Interval: 480 to < 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QTCB Interval: > 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QTCF Interval: 450 to 480 msec | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Maximum QTCF Interval: 480 to < 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum QTCF Interval: > 500 msec | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Max. QTC Interval Increase from BL: change ≥30 <60 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  QTC Interval Increase from BL: change ≥ 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Healthy Subjects: Maraviroc 150 mg twice a day (BID) co-administered with saquinavir 1,000 mg/ritonavir 100 mg twice a day (BID) for 7 days.
- Moderate Renal Impairment: Maraviroc 150 milligrams (mg) every 48 hours co-administered with saquinavir 1,000 mg/ritonavir 100 mg twice a day (BID) for 7 days.
- Severe Renal Impairment:: Maraviroc 300 mg single dose.
- ESRD: Dosing After Dialysis: Maraviroc 300 mg single dose one hour following completion of morning hemodialysis.
- ESRD: Dosing Before Dialysis: Maraviroc 300 mg single dose three hours prior to start of hemodialysis.
Arm/Group | Healthy Subjects | Mild Renal Impairment | Moderate Renal Impairment | Healthy Subjects: Single Dose | Severe Renal Impairment: | ESRD: Dosing After Dialysis | ESRD: Dosing Before Dialysis
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 6/6 | 6/6 | 1/6 | 3/6 | 2/6 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Subjects (N=6) | Mild Renal Impairment (N=6) | Moderate Renal Impairment (N=6) | Healthy Subjects: Single Dose (N=6) | Severe Renal Impairment: (N=6) | ESRD: Dosing After Dialysis (N=6) | ESRD: Dosing Before Dialysis (N=6)
conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 | 0 | 0 | 0 | 0 | 0
visual impairment (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
diarrhea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
flatulence (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
fatigue (General disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
sensation of foreign body (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
rhinitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
blood creatinine increased (Investigations) | 0 | 4 | 4 | 0 | 0 | 0 | 0
blood urea increased (Investigations) | 0 | 3 | 0 | 0 | 0 | 0 | 0
renal function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
headache (Nervous system disorders) | 2 | 3 | 1 | 0 | 0 | 0 | 0
paraesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
nocturia (Renal and urinary disorders) | 0 | 3 | 3 | 0 | 0 | 0 | 0
renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.